CLINICAL TRIAL: NCT06167603
Title: Exploring Brain Molecular Imaging and Blood Biomarkers in Subjects With Glucocerebrosidase Mutations: Toward a Precision Medicine Approach to Characterize Parkinson's Disease Clinical Trajectories
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: GR-2021-12373993
Record Dates: First submitted 2023-11-24; First posted 2023-12-12 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Hematologic Tests; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FDG-PET — Among other neuroimaging techniques, FDG-PET represents a unique tool to study the early metabolic alterations associated with neurodegeneration, both at the group and individual subject level.
Diagnostic Test: Blood test and clinical examination. — baseline, 12-months and 24 months.

SUMMARY:
Glucocerebrosidase (GBA) mutations are the most common risk factor for Parkinson's Disease (PD). GBA-related PD(GBA-PD) exhibits a more malignant phenotype as compared to no-carriers. Still, the mechanisms behind the increased malignancy in GBA-PD are not well understood. The definition of biomarkers able to stratify PD clinical trajectories in PD is therefore crucial to identify effective treatments and support diagnosis.The investigators will examine the role of GBA-mutations in accelerating a-synuclein (a-syn) and synaptic pathologies in PD by combining neuroimaging (positron emission tomography-PET), biochemical and clinical features. This will illuminate the pathophysiology underlying GBA-mutations in PD and identify biomarkers for the malignant PD phenotype. Also, the investigators will combine longitudinal clinical and imaging/biochemical features to define a prognostic algorithm for predicting disease faster progression in GBA-PD and monitoring disease trajectories in unaffected GBA carriers.

ELIGIBILITY:
Inclusion Criteria:

* PD diagnosis according to MDS-PD criteria and for GBA-PD group, presence of heterozygous GBA mutations;
* disease duration 3-7years.

Exclusion Criteria:

* other neurological or systemic diseases;
* presence of mutations in another PD gene;
* impossibility or unwillingness to perform FDG-PET.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients with and without GBA mutations and asymptomatic GBA mutation carriers, relatives of GBA-PD patients.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
FDG-PET to measure cerebral metabolism between Parkinson's subjects with a mutation in GBA gene (MP-GBA) compared to patients with idiopathic Parkinson's. | 3 years
  Differences in expression levels of posterior cerebral metabolism between Parkinson's patients with GBA mutation and idiopathic Parkinson's patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurological Institute Foundation Casimiro Mondino, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No